CLINICAL TRIAL: NCT05736406
Title: An Interventional, Multicenter, and International Phase 1/2, Light-dose-escalation Study to Investigate the Safety and Feasibility of Intraoperative Photodynamic Therapy (PDT) With Pentalafen® Drug and Heliance® Solution Device in Male and Female Patients 18 to 75 Years of Age With Grade IV Glioblastoma.
Brief Title: A Dose-escalation Clinical Study of Intraoperative Photodynamic Therapy of Glioblastoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hemerion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HTX-GBM-01; 2025-520563-41-00 (EU CTIS Number); 2025-A00107-42 (Other: ANSM)
Record Dates: First submitted 2023-02-08; First posted 2023-02-21 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Primary Glioblastoma
Keywords: Glioma; Glioblastoma; High Grade Glioma
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — 1-phenyl-3,3-dimethyltriazene; Aminolevulinic Acid

STUDY DESIGN:
Intervention Model Description: 3+3 model.The dose of light will be escalated in successive cohorts of patients. The starting dose is at 200 J/cm2. Enroll 3 patients at the first dose level and proceed to the next higher dose level with a cohort of 3 patients until at least 1 patient experiences a dose-limiting toxicity (DLT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- 200 J/cm^2 (Experimental): Patient will undergo intraoperative Photodynamic therapy at 200 J/cm^2
  Interventions: Combination Product: 5-ALA HCl intraoperative Photodynamic Therapy (PDT) at 200 J/cm^2
- 400 J/cm^2 (Experimental): Patient will undergo intraoperative Photodynamic therapy at 400 J/cm^2
  Interventions: Combination Product: 5-ALA HCl intraoperative Photodynamic Therapy (PDT) at 400 J/cm^2

INTERVENTIONS:
Combination Product: 5-ALA HCl intraoperative Photodynamic Therapy (PDT) at 200 J/cm^2 — 5-ALA HCl, 20 mg/kg, is orally administered 4-6 hours before the surgery. Then after resection of tumor tissue is judged maximal, the intraoperative PDT procedure is initiated at 200 J/cm^2.
  Other Names: Pentalafen®; 5-aminolevulinic acid hydrochloride; Heliance® Solution; 5-ALA PDT
  Arms: 200 J/cm^2
Combination Product: 5-ALA HCl intraoperative Photodynamic Therapy (PDT) at 400 J/cm^2 — 5-ALA HCl, 20 mg/kg, is orally administered 4-6 hours before the surgery. Then after resection of tumor tissue is judged maximal, the intraoperative PDT procedure is initiated at 400 J/cm^2.
  Other Names: Pentalafen®; 5-aminolevulinic acid hydrochloride; Heliance® Solution; 5-ALA PDT
  Arms: 400 J/cm^2

SUMMARY:
The primary objective of this clinical trial is to determine the safety and tolerability of two doses of light in intraoperative PDT added to standard of care; temozolomide-based chemotherapy in male and female patients aged 18 to 75 with newly diagnosed glioblastoma.

This treatment will be carried out in addition to the maximal surgical resection. Data collected during this trial will be used to design the upcoming pivotal study .

The study will utilize an independent Data and Safety Monitoring Board (iDSMB) that will review safety data to allow dose escalation.

DETAILED DESCRIPTION:
This study is a non randomized, open label, multicentercenter , phase 1/2 trial with a sequential enrollment in a 3+3 dose escalation design to establish the maximal tolerated dose of light (MTD).

The dose of light will be escalated in successive cohorts of patients until at least 1 patient experiences a dose-limiting toxicity (DLT).

A DLT is defined as any grade ≥ 3 Adverse Event (AE), or any relevant grade 2 AE of Central Nervous System or any Serious Adverse Events (SAEs) possibly, probably or definitively related to the intraoperative PDT (i.e., 5-aminolevulinic acid hydrochloride (5-ALA HCl) administration + brain cavity illumination), for which the onset date is within 28 days after the procedure, and where conservative therapy fails and surgical is required, according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

After dose escalation patient will be followed in the standard of care until visit at 6 months to evaluate the progression free survival.

ELIGIBILITY:
Inclusion criteria I01. Males or females must be between 18, or legal age of consent, and 75 years of age (both included) at the time of signing informed consent.

I02. Signed informed consent which includes compliance with requirements and restrictions listed in the informed consent.

I03. Newly diagnosed GBM, presumed on the basis of clinical and MRI criteria (intra-axial brain tumor with peripheral rim contrast enhancement).

I04. Karnofsky Performance Score ≥70 I05. Eligible for surgery. I06. Amenable to maximal tumor resection based on MRI. I07. Planned to receive SOC (i.e., Stupp Protocol) treatment after surgery. I08. Ability to take oral medications. I09. Tumor eligible to PDT procedure as validated by both investigator and sponsor based on pre-operative MRI data

Exclusion criteria

1.Medical conditions E01.

1. Patient with bifocal or multifocal disease, assessed on MR1I T1Gd enhanced.
2. Patient with tumor of deep location such as tumor involving the corpus callosum, the basal ganglia, the brain stem, or tumor involving the midline as assessed on MRI.
3. Patient with prior brain surgery other than stereotactic biopsy E02. Patient with Lynch syndrome E03. Patient with Li-Fraumeni syndrome E04. Debilitating cardiopulmonary disease, unstable Type 1 or Type 2 diabetes (treated or not) E05. History or current condition of another malignancy (excluding basal cell carcinoma, or E05. carcinoma in-situ) unless treated and off all active therapy for more than 5 years E06. Clinically significant abnormal ECG results, including a corrected QT interval QTc > 480 ms E07. Creatinine clearance < 60 mL/min E08. Severe hepatic impairment (bilirubin > 1.5 x the upper limit of normal [ULN] or alkaline phosphatase or transaminases (AST, ALT) > 2.5 x ULN) E09. Known allergic reactions to silicone E10. Known allergic reactions or hypersensitivity to egg, soya, or peanut proteins.

E11. Febrile illness

Contraindication

E12. Contraindication to 5-ALA HCl administration, including:

1. Porphyria
2. Taking photosensitizing drugs 24 hours before and 14 days after the administration of Pentalafen® including but not limited to: St. John's wort, griseofulvin, thiazide diuretics, sulfonylureas, phenothiazines, sulphonamides, quinolones and tetracyclines, and topical preparations containing ALA (See Section 6.10)
3. Inability to suspend a long-term hepatotoxic treatment (such as, but not limited to diclofenac, fenofibrate, carbamazepine) for 24 hours after 5-ALA HCl intake E13. Contraindication to MRI examination (e.g., MRI-incompatible pacemaker) E14. Treatment with another investigational drug or intervention within 30 days prior to or during the entire study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Maximal Tolerated Dose (MDT) of light for Photodynamic Therapy | 4 weeks after intervention
  Evaluation of Dose Limiting Toxicities (DLT) to define MDT

SECONDARY OUTCOMES:
Treatment response / Progression-free survival (PFS) | Up to 6 months after intervention
  MRI imaging and RANO criteria
Number of Adverse Events and Serious Adverse Events (Safety and Tolerability) | 6 months
  Global clinical safety data of 5-ALA HCl Intraoperative PDT

OTHER OUTCOMES:
Usability of the Heliance® Solution in the operating room | During Procedure
  Score of usability calculated from usefulness, ease of use, ease of learning and satisfaction/intention of use measures

CONTACTS AND LOCATIONS:
Overall Officials: Jan Drappatz, MD, Principal Investigator — UPMC Presbyterian Shadyside Hospital, Pittsburgh, PA
Locations (2):
- UPMC Hillman Cancer center, Pittsburgh, Pennsylvania, United States
- CHU De Lille, Hôpital Roger Salengro, Lille, France

IPD SHARING:
Plan to Share IPD: No